CLINICAL TRIAL: NCT06639113
Title: Evaluation of the Safety of a Change of Practice in the Administration of Oral Medication During Hospitalisation: From Administration by the Nurse to Supervision of Self-administration of Medication in the Locomotor and Polyvalent Rehabilitation Department of the Valenciennes Hospital Centre.
Brief Title: From Administration of Oral Medicines by Nurses to Controlled Self-administration: Impact on Safety of Administration During Hospitalisation
Acronym: AUTOGESTMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02-04
Record Dates: First submitted 2024-09-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Self Administration
Keywords: Rehabilitation; Self-management of medication; Administration; Autonomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self administration of medication by the patient (Experimental): Self administration of medication by the patient
  Interventions: Behavioral: Self-administration medicines
- Administration of medication by the nurses (No Intervention): Administration of medication by the nurses during medication administration rounds

INTERVENTIONS:
Behavioral: Self-administration medicines — Management of drugs' administration by the patient
  Arms: Self administration of medication by the patient

SUMMARY:
Medication administration practices during patient hospital stay tend to improve patient autonomy. Several studies have concluded that self-administration of medication programs in hospital centers have a beneficial effect on patients' knowledge of their medications, their compliance and the safety of administration. Nevertheless, few studies have been carried out in France on this subject. The aim of this study is to evaluate the impact of the change of nurses administration practices from the administration of each drugs to supervision of self-administration by the patient under a self-administration program.

ELIGIBILITY:
Inclusion Criteria:

* Care in the rehabilitation unit of Hospital in Valenciennes, France
* Patient with a planned stay of 7 days or more
* Patient on chronic treatment before admission to hospital ;
* Patients taking their treatment alone at home;

Exclusion Criteria:

* Age < 18 years old
* Patients with poor compliance
* No chronic treatment
* Unstable disease
* Major cognitive, memory or depressive disorders
* Swallowing disorders
* Prehension problems
* Patient under legal protection
* Patient under guardianship or curatorship
* Patient included in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Total number of oral medication administration errors in self-administered patients | After 7 days of self-administration
  Total number of oral medication administration errors in self-administered patients
Total number of oral medication administration errors in patients receiving administration by nurses | After 7 days of administration by nurses
  Total number of oral medication administration errors in patients receiving administration by nurses

SECONDARY OUTCOMES:
Medication compliance in self-managed patients | At the beginning of the study
  Medication compliance is assessed using the questionnaire "Evaluation of medication compliance" provided by the French health insurance system.
  This questionnaire consists of 6 questions with "yes" or "no" answers. Each "no" answer is worth 1 point, each "yes" answer is worth 0 points. A patient with poor medication compliance will have a score of 3 or less.
Medication compliance in self-managed patients | 15 days after hospital discharge for self-managed patients
  Medication compliance is assessed using the questionnaire "Evaluation of medication compliance" provided by the French health insurance system.
  This questionnaire consists of 6 questions with "yes" or "no" answers. Each "no" answer is worth 1 point, each "yes" answer is worth 0 points. A patient with poor medication compliance will have a score of 3 or less.
Patient satisfaction with self-administration of oral medication | Within 24 hours of discharge from hospital
  Patient satisfaction was assessed using a questionnaire designed by the investigator, consisting of 9 questions giving a total of 45 points.
  The higher the total, the higher the level of satisfaction.
Care staff satisfaction with self-administration | 6 months after the beginning of the study
  Care staff satisfaction was assessed using a questionnaire designed by the investigator, consisting of 4 questions totalling 20 points.
  The higher the total, the higher the level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Quentin HIVER, PH, Principal Investigator — Centre Hospitalier de Valenciennes
Locations (1):
- CH Valenciennes, Valenciennes, France

IPD SHARING:
Plan to Share IPD: No